CLINICAL TRIAL: NCT02625025
Title: Low vs Standard Pneumoperitoneum Pressure During Single Port Access Laparoscopic for Adnexal Pathology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPALPression
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Adnexal Benign Pathology

ARMS (2):
- Low pression pneumoperitoneum (Experimental): Patients undergoing Single Port Access Laparoscopy for benign adnexal pathology with use of Low Pression Pneumoperitoneum (8 mm Hg)
  Interventions: Procedure: Low pression pneumoperitoneum; Procedure: Single Port Access Laparoscopy
- Standard pression pneumoperitoneum (Experimental): Patients undergoing Single Port Access Laparoscopy for benign adnexal pathology with use of Standard Pression Pneumoperitoneum (12 mm Hg)
  Interventions: Procedure: Standard Pression Pneumoperitoneum; Procedure: Single Port Access Laparoscopy

INTERVENTIONS:
Procedure: Low pression pneumoperitoneum — Pneumoperitoneum will be obtained by infusing carbon dioxide to distend the peritoneal cavity.
  Intra-abdominal pressure will be maintained at 8 mm Hg during pneumoperitoneum creation and insertion of trocars.
  Arms: Low pression pneumoperitoneum
Procedure: Standard Pression Pneumoperitoneum — Pneumoperitoneum will be obtained by infusing carbon dioxide to distend the peritoneal cavity.
  Intra-abdominal pressure will be maintained at 12 mm Hg during pneumoperitoneum creation and insertion of trocars.
  Arms: Standard pression pneumoperitoneum
Procedure: Single Port Access Laparoscopy — Laparoscopy surgery with use of only one incision of 2 cm in the umbilicus in order to threat benign adnexal pathology

SUMMARY:
During laparoscopy pneumoperitoneum creates the necessary space in which to perform the operation. Growing evidence in general surgery has shown that reduction of intra-abdominal pressure during laparoscopy is related to improved postoperative outcomes, decreased pain perception, length of hospital stay, and analgesic rescue dosage in patients undergoing minimally invasive procedures using low pneumoperitoneum pressure (LPP) compared with standard pneumoperitoneum pressure (SPP). Aim of the study is to demonstrate the safety and feasibility of LPP during performance of Single Port Access Laparoscopy for benign adnexal pathologies.

ELIGIBILITY:
Inclusion Criteria:

* patients 18- 45 years old
* elective laparoscopic operation
* informed consent

Exclusion Criteria:

* BMI > 30 kg/cm2
* pregnancy
* converting to laparotomy
* malignant disease
* unable or unwilling to give written consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measured on a VAS scale | 6 hours
  Experienced pain over the last six hours measured on a VAS scale

SECONDARY OUTCOMES:
Operation time | 0 hours after the operation
  Operating time in minutes.
Blood loss in ml | 0 hours after the operation
  Estimated blood loss in ml.
Complications | Two months
  Complications during surgery and late complications.
Shoulder tip pain measured on a VAS scale | 24 hours
  Experienced shoulder tip pain over the last 24 hours measured on a VAS scale.
Postoperative pain measured on a VAS scale | 24 hours
  Experienced pain over the last 24 hours measured on a VAS scale.